CLINICAL TRIAL: NCT02751190
Title: Chronic Pain After Groin Hernia Repair, Impact of Method of Surgery
Brief Title: Chronic Pain After Groin Hernia Repair
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: JLL-468171
Record Dates: First submitted 2016-04-08; First posted 2016-04-26 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2016-04

CONDITIONS: Hernia, Inguinal; Hernia, Femoral
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral | interventions — tetraethylpyrazine; Wound Healing; tetra-4-amidinophenoxypropane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Totally ExtraPeritoneal (TEP) repair
Procedure: TransAbdominal PrePeritoneal (TAPP) repair
Procedure: Open anterior mesh repair
  Other Names: Lichtenstein repair
Procedure: Open Anterior Non Mesh
  Other Names: McVay; Bassani; Shouldice; Marcy
Procedure: Combined anterior and posterior repair
  Other Names: Plug; Prolene Hernis System (PHS); Onstep; TransInguinalPrePeritoneal repair (TIPP)
Procedure: Open preperitoneal mesh repair
  Other Names: Nyhus; Stoppa; Rives

SUMMARY:
In the present study the investigators aimed to investigate the relationship between surgical methods and chronic pain in over 20 000 patients who underwent groin hernia repair in Sweden

DETAILED DESCRIPTION:
The Swedish Hernia Register (SHR) covers more than 98% of all groin hernia repairs in Sweden. Approximately 16.000 hernia repairs is performed annually. All patients are identified by the Swedish personal identification number (PIN), which is assigned at birth and used in virtually all contacts with Swedish healthcare and authorities.

All variables in the SHR are collected prospectively at the time of surgery, reported by the surgeon. Variables collected are numerous and contain among else age, gender, method of repair, anaesthesia type, hernia anatomy, recurrent or primary repair, sliding hernia, handling of the hernia sac, resident or consultant surgeon, annual surgeon volume, and type of unit.

A detailed variable list is found at the Swedish National Board of Welfare website (http://www.socialstyrelsen.se/register/registerservice/nationellakvalitetsregister/svensktbrackregister-nationell) Variables are validated thru annual validation of 10% of participating units where register data are checked against chart review made on a randomized sample of patients and units.

Patient can be registered more than once and be followed in time, which is possible by using the PIN.

Preoperative pain is not registered.

Starting 2013, a questionnaire regarding Patient Reported Outcome Measure (PROM) is sent to all patients having an groin hernia repair from September 2012 until December 2014. Patients are identified in the SHR and postal addresses obtained through the register of the whole population, using the PIN.

Patients were sent a short form of Inguinal Pain Questionnaire (IPQ). IPQ is a validated pain questionnaire, specifically designed for groin hernia repair. The key question sent were " Grade the pain you felt in the operated groin the last week". Patients then answered in a 7 grades scale, where pain was correlated to if it could be ignored and to what extent it limited activities of daily life.

The questionnaire could be answered on regular paper or through a web questionnaire. One reminder was sent if no answer was collected within 1 month

The surgical methods were divided in 5 groups. Total ExtraPeritoneal (TEP) (Reference group), TransAbdominal PrePeritoneal (TAPP), Open anterior mesh technique (OAM i.e Lichtenstien), Open anterior non mesh ( ONM i.e Shouldice, McVay, Bassini), Combined Anterior end posterior Techniques (CAP i.e. Plug, Prolene Hernia System, Onestep), and Open Preperitoneal Mesh Techniques (OPT).

The method of surgery and other variables at index surgery for each individual patient was derived from the SHR through the PIN.

Using data from SHR. Multivariate analysis and propensity score matching will be used for analysis. Adjustments is made for all known and possible confounders such as age (above or below median age), gender, primary or recurrent hernia, emergent or electively operated, ASA class (≤2/>2),mesh weight (light (≤50g/m2) or heavy (> 50g/m2)), resident or consultant surgeon, annual surgeon volume (≤25/>25), hernia anatomy (femoral/medial/lateral- combined hernias considered as lateral), per or postoperative complication yes/no (hematoma, severe pain, infection and other complications), handling of the hernia sac (divided excised or invaginated) and type of hospital and others.

Missing data on different variables is managed by exclusion or imputation.

Adverse events such as preoperative complication is reported by the surgeon, and postoperative complications are detected by registry administrator at the surgical site by chart review 30 days postoperatively.

A reliability test (test-retest) is made on a random sample of patients 30 days apart.

A non responder analysis is conducted to asses wether patients not responding on the primary questionnaire differs from the responders according to perceived pain. This is done by randomly select patients to conduct a telephone interview.

Power calculations is based on the assumption of 75% response rate (0.75x30.000)= 22.500. Of these approximately 15% TEP=3375. Of TEP approximately 50% is done bilaterally, which is excluded from this study. Assuming a difference in pain of 4% in favor of TEP, it is needed more than 1200 patients in the TEP group to detect these differences, considered clinically meaningful.

ELIGIBILITY:
Inclusion criteria:

* Unilateral, elective, groin hernia repair

Exclusion criteria:

* Bilateral hernia repair
* Emergent repair (<24h of duration with signs of incarceration)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients registered in the Swedish hernia surgery.
Sampling Method: Probability Sample
Enrollment: 24607 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Chronic post herniorraphy pain | 1 year
  A IPQ score of > 3. Pain, which could not be ignored and affected concentration on activities and leisure activities

SECONDARY OUTCOMES:
Reoperation for recurrence | Up to 4 years from primary surgery
  Reoperation for recurrence in the same groin (all types of groin hernias)

CONTACTS AND LOCATIONS:
Overall Officials: Pär Nordin, MD.Ph.D, Principal Investigator — Umea University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900
- [Background] Nilsson E, Haapaniemi S. Assessing the quality of hernia repair. In: Fitzgibbons RJ, Nyhus LM, eds. Hernia. Philadelphia: Lippincott Williams and Wilkins, 2002:567-73.